CLINICAL TRIAL: NCT00983086
Title: Effects of Consumption of Orange Juice on Vascular Protection and Immune Function: Clinical Study on the Specific Contribution of Citrus Flavanones
Acronym: FLORIDE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Patrick Lacarin, CHU Clermont-Ferrand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0059
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Volunteers
Keywords: Flavanones and vascular function

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Flavanones of orange juice — The main objective of this study is to evaluate, in healthy volunteers with young children (50 and 65) and slightly overweight according to their usual diet, the effects of single dose (in postprandial period) and made repeated orange juice or orange flavanones purified on vascular function. The selection criteria for age and weight should, within a healthy population to select individuals who exhibit cardiovascular risk factors, and thus for which it should be a priori easier to identify a beneficial effect of dietary factors on the parameters associated with cardiovascular risk.

SUMMARY:
Epidemiological studies have firmly established the health effects of high intakes of fruits and vegetables and in particular in regards to the prevention of cardiovascular diseases. Citrus fruits are the most widely consumed throughout the world, mainly as juice. Citrus fruits are rich in vitamin C but also in various plant micronutrients which are the most abundant polyphenols. Several in vitro studies and animal models suggest that the polyphenols of citrus are involved in the protective effects of citrus vis-à-vis the cardiovascular diseases. However, profits in health associated with taking these polyphenols are unknown and so far no clinical studies have been conducted to determine the contribution of polyphenols of citrus in this protection.

The main objectives of this project are (1) to characterize the effects of single dose and made repeated consumption of orange juice on vascular protection and the immune response and (2) to assess the specific role of polyphenols present in citrus fruits in this protection. To do this the investigators will conduct a clinical study, randomized and crossover, among healthy men 50 to 65 years that are slightly overweight. These volunteers, who continue to follow their usual diet, should consume daily for 4 weeks (1) orange juice or (2) an isocaloric control beverage or (3) the same drink spiked with a dose of polyphenols similar to that given by orange juice.

DETAILED DESCRIPTION:
Clinical study, randomized, crossover, double-blind in healthy men 50 to 65 years who are slightly overweight.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Age: 50 to 65 inclusive
* Body mass index of 25 to 30 kg / m² (inclusive

Exclusion Criteria:

* Hypertriglyceridemia or known hypercholesterolemia, treated or not
* Serology HIV and / or HCV positive

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Determine the effects of repeated consumption of orange juice or purified flavanones in immune function | after consumption of orange juice

SECONDARY OUTCOMES:
Measuring the impact of consumption of orange juice or purified flavanones on acid-base balance | after consumption of orange juice
Evaluate the effects of chronic consumption of orange juice or purified flavanones on gene expression by a global transcriptomic approach in mononuclear cells from peripheral blood | after consumption of orange juice

CONTACTS AND LOCATIONS:
Overall Officials: Claude Dubray, PU PH, Principal Investigator — University Hospital, Clermont-Ferrand

REFERENCES:
- [Derived] Milenkovic D, Deval C, Dubray C, Mazur A, Morand C. Hesperidin displays relevant role in the nutrigenomic effect of orange juice on blood leukocytes in human volunteers: a randomized controlled cross-over study. PLoS One. 2011;6(11):e26669. doi: 10.1371/journal.pone.0026669. Epub 2011 Nov 16. PMID 22110589
- [Derived] Morand C, Dubray C, Milenkovic D, Lioger D, Martin JF, Scalbert A, Mazur A. Hesperidin contributes to the vascular protective effects of orange juice: a randomized crossover study in healthy volunteers. Am J Clin Nutr. 2011 Jan;93(1):73-80. doi: 10.3945/ajcn.110.004945. Epub 2010 Nov 10. PMID 21068346